CLINICAL TRIAL: NCT04887792
Title: A Randomized Controlled Trial of Acetazolamide for Patients With Treatment Resistant Schizophrenia
Brief Title: Acetazolamide for Treatment Resistant Schizophrenia
Acronym: APTS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vishwajit Nimgaonkar, MD PhD (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Vishwajit Nimgaonkar, MD PhD, Professor of Psychiatry and Human Genetics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20010237
Record Dates: First submitted 2020-12-15; First posted 2021-05-14 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia; Schizo Affective Disorder
Keywords: Schizophrenia; Schizo Affective Disorder; acetazolamide
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: This study will be a randomized placebo-controlled sequential parallel comparison design (SPCD).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care providers, Investigators and assessors will all be blinded. Study staff responsible for randomization will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetazolamide (Active Comparator): acetazolamide capsules
  Interventions: Drug: Acetazolamide
- Placebo (Active Comparator): Identical gelatin capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — ACZ 250 mg/day in gelatin capsules will be administered initially and increased over 7-10 days to 2g/day.
  Other Names: Diamox
  Arms: Acetazolamide
Drug: Placebo — Identical gelatin capsules will be prepared by filling with inert excipients.
  Arms: Placebo

SUMMARY:
This is a double blind adjunctive randomized controlled trial for schizophrenia using acetazolamide.

DETAILED DESCRIPTION:
Schizophrenia (SZ) afflicts over 21 million people worldwide. Persons with SZ have a 10% suicide rate and their lifespan is curtailed by over 25 years. There is an urgent need for efficacious antipsychotic drugs (APDs), particularly, second line drugs, because only 30-40% of APD-treated patients attain remission and 30% of patients show little or no response. Currently, Clozapine is the only reliable second line APD, but it can cause serious blood dyscrasias. To fill the void, the investigators have conducted systematic reviews of prior data and in silico searches. In a prior double-blind crossover randomized placebo-controlled trial (RCT), adjunctive Acetazolamide (ACZ) caused ~20% improvement in positive and negative symptom scores when added to APDs among partially-responsive patients with SZ (ACZ 2G/day). No patients dropped out. The RCT is supported by several other open trials. ACZ also reduces weight, thus it could combat weight gain, a common APD side effect. Independently, our systematic in silico strategy based on protein networks and gene expression profiles also identified Acetazolamide (ACZ) as a repurposable drug for SZ.

ACZ crosses the blood-brain barrier. It is used to treat CNS diseases such as refractory seizures and idiopathic intracranial hypertension. Used for over 50 years, its side effects (SE) and adverse effects (AE) are well known and are manageable. It is a potent, specific inhibitor of carbonic anhydrase (CA), which catalyzes the conversion of CO2 to HCO3- and H+. CA is localized to pre-synaptic terminals and glial cells. It modulates GABAergic excitation, long-term synaptic transformation, attentional gating of memory storage and cerebrospinal fluid formation. Post-mortem brain and serological studies show raised CA levels in patients with psychotic/mood disorders. Several APDs also inhibit CA. The investigators thus postulate brain CA inhibition as the therapeutic target for ACZ in SZ.

The investigators propose a double-blind, crossover RCT for SZ using adjunctive ACZ. To maximize the risk/benefit ratio, the investigators will enroll inpatients and outpatients with treatment resistant SZ (trSZ) who meet defined criteria (N=60 RCT completers). ACZ or placebo will be added to prescribed APDs for 8 weeks utilizing the Sequential Parallel Comparison Design to maximize power. The investigators have extensive experience with RCTs. The investigators will ensure timely recruitment by approaching a large group of patients we serve, across 2 sites. If ACZ is beneficial, in future studies the investigators will pursue its implementation for trSZ, and seek variables associated with treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Both genders, ages 18-55 years (older patients may not tolerate high ACZ dose).
* PANSS total score > 60 and Score > 4 on one or more items of the 'positive' syndrome items (P1-P7), following treatment at therapeutic doses for 6 weeks with different APDs on 2 occasions.
* Stable dose of antipsychotic drug (APD) for > 1 month, continued throughout the study.
* Not participating in another randomized controlled clinical trial (RCT).

Exclusion Criteria:

* Substance abuse in the past month/dependence past 6 months with the exception of methadone prescribed for opiate withdrawal.
* History or current medical/neurological illnesses that may lead to unstable course, e.g., epilepsy.
* Pregnancy.
* Acetazolamide (ACZ) contraindications: hypersensitivity to ACZ; history of renal hyperchloremic acidosis; Addison's disease/adrenal failure; chronic closed angle-closure glaucoma.
* Current or prior treatment with ACZ or history of hypersensitivity to ACZ.
* Intellectual disability as defined in DSM 5.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in positive symptoms | 24 weeks
  Clinical Severity as determined by the Positive and Negative Syndrome Scale (PANSS) positive symptom subscale. The PANSS is a standardized, clinical interview that rates the presence and severity of positive and negative symptoms, as well as general psychopathology for people with schizophrenia within the past week. Symptom severity for each item is rated according to which anchoring points in the 7-point scale (1 = absent; 7 = extreme) best describe the presentation of the symptom. 7 Items, (minimum score = 7, maximum score = 49)

SECONDARY OUTCOMES:
Clinical Severity | 24 weeks
  Clinical Severity as determined by the Positive and Negative Syndrome Scale (PANSS) positive symptom subscale. The PANSS is a standardized, clinical interview that rates the presence and severity of positive and negative symptoms, as well as general psychopathology for people with schizophrenia within the past week. Symptom severity for each item is rated according to which anchoring points in the 7-point scale (1 = absent; 7 = extreme) best describe the presentation of the symptom. 30 Items, (minimum score = 7, maximum score = 210)
Clinical Severity | 24 weeks
  Clinical Severity as determined by the Positive and Negative Syndrome Scale (PANSS) positive symptom subscale. The PANSS is a standardized, clinical interview that rates the presence and severity of positive and negative symptoms, as well as general psychopathology for people with schizophrenia within the past week. Symptom severity for each item is rated according to which anchoring points in the 7-point scale (1 = absent; 7 = extreme) best describe the presentation of the symptom. 7 Items, (minimum score = 7, maximum score = 49)
Cognition | 24 weeks
  Trail Making Test (TMT) 86: This test estimates attention, working memory and executive function.
Clinical Severity | 24 weeks
  "Clinical Global Impression - Severity" (CGI-S). The CGI-S is a 7-point scale that rates the severity of the patient's illness at the time of assessment. The minimum score is 1 and the maximum score is 100. Scores which are lower in value indicate greater severity of illness. Higher scores indicate less severe illness.
Social Function | 24 weeks
  "Sheehan's Disability Scale" (SDS). The SDS is a self-report is a self-report tool that assesses functional impairment in work/school, social and family life with a 10-point visual analogue scale. The minimum score is 0 and the maximum score is 10. Scores which are lower in value indicate better outcomes with less disability. Higher scores indicate more severe illness with greater disability.
Global Assessment of Function | 24 weeks
  "Global Assessment of Function" (GAF). The GAF is an assessor reporting tool that assesses level of functioning on a 1 to 100 point scale. The minimum score is 1 and the maximum score is 100. Scores which are higher in value indicate better outcomes with less disability. Lower scores indicate more severe illness with greater disability.
Measure of satisfaction with one's Quality of Life (Quality of Life Scale/QOLS) | 24 weeks
  The QOLS was originally a 15-item instrument that measured five conceptual domains of quality of life: material and physical well-being, relationships with other people, social, community and civic activities, personal development and fulfillment, and recreation. After descriptive research that queried persons with chronic illness on their perceptions of quality of life, the instrument was expanded to include one more item: Independence, the ability to do for yourself. Thus, the QOLS in its present format contains 16 items.
  The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112. The QOLS scores are summed so that a higher score indicates higher quality of life. Average total score for healthy populations is about 90.
Socio-Economic Status | 24 weeks
  We will use a composite measure of educational attainment and pretax family (household) income based on the Hollingshead Redlich 4-factor index.
  The Hollingshead Four Factor Index of Socioeconomic Status is a survey designed to measure social status of an individual based on four domains: marital status, retired/employed status, educational attainment, and occupational prestige. The participant's education code is obtained education code is rated on a 7-point scale that lists highest grade completed. The participant's occupational code is rated on a 9-point scale.
  SES=0.5X education score+0.3Xincome score+ 0.3X occupation score.
Side Effects | 24 weeks
  We will make a list of side effects for CGY noted in the Drug Formulary. This list will be a comprehensive listing of possible side effects by body system, grading both the frequency and severity of the symptoms.
  Frequency (days per week): Severity:
  0 = Absent
  1. = 1-2 days 1 = mild, does not interfere with functioning
  2. = 3-4 days 2 = moderate, some interference with functioning
  3. = 5-7 days 3 = severe, functioning is significantly impaired
  Frequency scores can range from 0 to 3, with higher scores equaling higher frequency.
  Severity scores can range from 1 to 3, with higher scores equaling greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, M.D., Ph.D., Principal Investigator — University of Pittsburgh
Locations (2):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States
- St John's Medical College Hospital, Bangalore, India

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared.